CLINICAL TRIAL: NCT00053911
Title: Randomized And Multicentric Phase III Study Evaluating The Benefit By Using A Chemotherapy With FEC 100 And Docetaxel In Non Metastatic Breast Cancer Which Has Relapsed After A Conservative Surgery
Brief Title: Combination Chemotherapy Compared With Observation After Surgery in Treating Women With Relapsed Nonmetastatic Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: PACS03; FRE-FNCLCC-PACS-03/003; EU-20237
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Cyclophosphamide; Docetaxel; Epirubicin; Fluorouracil; Goserelin; Tamoxifen; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: anastrozole
Drug: cyclophosphamide
Drug: docetaxel
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: goserelin acetate
Drug: tamoxifen citrate
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug, and giving them after surgery, may kill any remaining tumor cells following surgery. It is not yet known whether combination chemotherapy is more effective than observation in treating relapsed nonmetastatic breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with that of observation in treating women who have undergone surgery for relapsed nonmetastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of adjuvant cyclophosphamide, epirubicin, and fluorouracil vs observation, in terms of disease-free 5-year survival, in women who have undergone resection for relapsed nonmetastatic breast cancer after initial conservative surgery.
* Compare the overall survival of women treated with these regimens.
* Determine the tolerance of these women to the chemotherapy regimen.
* Correlate prognostic factors of survival with efficacy of the chemotherapy regimen in these women.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to menopausal status and participating center. Patients are randomized to 1 of 2 treatment arms. Study begins within 42 days after resection of recurrent disease.

* Arm I: Patients receive fluorouracil IV over 1 hour, epirubicin IV over 1 hour, and cyclophosphamide IV over 1 hour on day 1. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive docetaxel IV over 1 hour on day 1. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients are examined on days 1 and 63.

Patients who are hormone receptor positive also receive one of the following hormonal therapy regimens, depending on menopausal status:

* Oral tamoxifen daily for 5 years
* Oral tamoxifen daily for 5 years and oral luteinizing hormone-releasing hormone (LHRH) agonist therapy (e.g., goserelin) for 3 years
* Oral LHRH agonist therapy (e.g., goserelin) for 3 years
* Oral antiaromatase therapy (e.g., anastrozole) for 5 years Patients also undergo radiotherapy and may also undergo second complete resection.

Patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 370 patients (185 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * No contralateral breast cancer
* Local tumor recurrence more than 6 months after conservative surgery
* Complete or conservative resection of the recurrent tumor NOTE: Initial complete surgical resection not allowed
* No local inflammatory disease or disease that is not amenable to complete surgical resection
* No positive axillary lymph nodes
* No distant metastases, including subclavicular lymph nodes
* Hormone receptor status:

  * Hormone receptor status known

PATIENT CHARACTERISTICS:

Age

* 18 to 65

Sex

* Female

Menopausal status

* Menopausal status known

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* Transaminases no greater than 1.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* No chronic hepatitis B
* No active hepatitis C

Renal

* Not specified

Cardiovascular

* Cardiac function normal by echocardiogram or isotopes

Other

* No contraindications to anthracyclines such as any of the following:

  * Prior doxorubicin over 300 mg/m^2
  * Prior epirubicin over 600 mg/m^2
  * Prior mitoxantrone over 90 mg/m^2
* No other invasive malignancy
* No chronic somatic or psychiatric condition that would preclude study participation
* No familial, social, geographic, or psychological reason that would preclude study participation
* Not pregnant
* Fertile patients must use effective contraception
* HIV negative
* CA 153 no greater than 2 times ULN

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Patient Characteristics-Other
* No prior neoadjuvant chemotherapy

Endocrine therapy

* No prior neoadjuvant hormonal therapy

Radiotherapy

* No prior neoadjuvant radiotherapy

Surgery

* See Disease Characteristics
* At least 41 days since prior surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-11; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of the disease free survival | 5 years

SECONDARY OUTCOMES:
Evaluation of the overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Romieu, MD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (26):
- France (26):
  - Clinique Claude Bernard, Albi
  - Centre Paul Papin, Angers
  - Centre Hospitalier d'Annecy, Annecy
  - Institut Sainte Catherine, Avignon
  - Institut Bergonie, Bordeaux
  - C.H. Bourg En Bresse, Bourg-en-Bresse
  - CHU Hopital A. Morvan, Brest
  - Centre Hospitalier General, Brivé
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Compiegne, Compiègne
  - Clinique du Petit Colmouilins, Harfleur
  - Centre Oscar Lambret, Lille
  - Institut J. Paoli and I. Calmettes, Marseille
  - Hopital Notre-Dame de Bon Secours, Metz
  - C.H. General Andre Boulloche, Montbéliard
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Clinique Saint - Pierre, Perpignan
  - Centre Eugene Marquis, Rennes
  - Clinique Armoricaine De Radiologie, Saint Brieux
  - Polyclinique de L'Ormeau, Tarbes
  - Institut Claudius Regaud, Toulouse
  - Hopital J. Ducuing, Toulouse
  - Institut Gustave Roussy, Villejuif